CLINICAL TRIAL: NCT00627666
Title: Unrelated Donor Hematopoietic Stem Cell Transplantation After Nonmyeloablative Conditioning For Patients With Hematological Malignancies
Brief Title: Donor Stem Cell Transplant After Busulfan, Fludarabine, and Antithymocyte Globulin in Treating Patients With Hematological Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000583220; AMC-UUCM-2003-0207
Record Dates: First submitted 2008-02-29; First posted 2008-03-03 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2009-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; acute lymphocytic leukemia; secondary acute myeloid leukemia; acute undifferentiated leukemia; mast cell leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; chronic myelomonocytic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Leukemia, Mast-Cell; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Chronic; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Anemia, Refractory, with Excess of Blasts | interventions — Antilymphocyte Serum; Busulfan; fludarabine phosphate; Leucovorin; Methotrexate

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: fludarabine phosphate
Drug: leucovorin calcium
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor bone marrow stem cell transplant helps stop the growth of cancer cells. Chemotherapy and antithymocyte globulin stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and methotrexate after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving donor stem cell transplant together with busulfan, fludarabine, and antithymocyte globulin works in treating patients with hematological cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate whether unrelated donor hematopoietic stem cell transplantation using a nonmyeloablative conditioning regimen comprising busulfan, fludarabine phosphate, and anti-thymocyte globulin can reduce treatment-related mortality in patients with hematologic malignancies.
* To investigate whether this regimen can be sufficiently immunosuppressive to enable engraftment of HLA-matched unrelated hematopoietic stem cells.

OUTLINE: This is a multicenter study.

Prior to receiving the conditioning chemotherapy regimen, all patients with acute leukemia, chronic myelogenous leukemia (CML), and high-risk myelodysplastic syndromes (chronic myelomonocytic leukemia, atypical CML, and refractory anemia with excess blasts) receive one dose of intrathecal (IT) methotrexate. These patients also receive leucovorin calcium IV or orally 4 hours after IT methotrexate and every 6 hours for a total of 8 doses.

* Nonmyeloablative conditioning regimen: Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -2, busulfan IV over 3 hours on days -7 to -6, anti-thymocyte globulin IV over 4 hours on days -4 to -2.
* Allogeneic bone marrow stem cell transplantation (SCT): Patients undergo allogeneic bone marrow SCT on day 0.
* Graft-versus-host-disease (GVHD) prophylaxis: Patients receive cyclosporine (CSA) IV over 2-4 hours every 12 hours starting on day -1 and continuing until day 180 (CSA can be given orally every 12 hours once oral medication can be tolerated) and methotrexate IV on days 1, 3 , 6 , and 11.

Once blood counts recover, patients with acute leukemia or CML in blast crisis resume IT methotrexate once every 2 weeks for a total of 3 doses. Patients also receive leucovorin calcium IV or orally 4 hours after IT methotrexate and then every 6 hours for a total of 8 doses.

Patients are followed for at least 10 years after SCT.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any 1 of the following:

  * Acute leukemia
  * Chronic myelogenous leukemia
  * Myelodysplastic syndromes
* Must have an unrelated donor available who is matched for HLA-A and -B by serology and for DRB1 by molecular typing

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Bilirubin < 3.0 mg/dL
* Creatinine < 2.0 mg/dL
* AST and ALT < 3 times the upper limit of normal
* Not pregnant or nursing
* Ejection fraction ≥ 45% by MUGA scan or ECHO
* No major illness or organ failure
* No severe psychiatric disorder or mental deficiency that makes compliance with the treatment unlikely and informed consent impossible

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2003-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Treatment-related mortality
Engraftment

SECONDARY OUTCOMES:
Regimen-related toxicities
Graft-versus-host-disease
Relapse
Overall survival
Failure-free survival
100-day transplant-related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo H. Lee, MD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center - University of Ulsan College of Medicine, Seoul, South Korea

REFERENCES:
- [Result] Lee KH, Choi SJ, Lee JH, Lee JH, Kim DY, Seol M, Lee YS, Kang YA, Jeon M, Yun SC, Joo YD, Lee WS, Kang MJ, Kim H, Park JH, Bae SH, Ryoo HM, Kim MK, Hyun MS. Clinical effect of reduced-intensity conditioning regimen containing antithymocyte globulin for hematopoietic cell transplantation from unrelated-donors. Am J Hematol. 2011 May;86(5):399-405. doi: 10.1002/ajh.21989. PMID 21523798